CLINICAL TRIAL: NCT02673346
Title: Assessing Tobacco Use and Treatment Preferences Among Alaska Yukon-Kuskokwim Health Corporation Employees
Brief Title: Employee Wellness Survey
Acronym: Wellness
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Yukon Kuskokwim Health Corporation (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Other Study IDs: 14-007166
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- employees: YKHC employees

SUMMARY:
The aims of this study are 1) To assess the prevalence of tobacco use and cessation treatment preferences among YKHC employees, 2) To assess employee's current levels of perceived stress, engagement in physical activity, and feelings of resiliency to inform future tobacco cessation interventions, and to examine the relationship between these factors and tobacco use, and 3) To assess YKHC employees' perceptions and opinions of the hospital's current workplace tobacco policy and expansion of these regulations to all YKHC properties.

DETAILED DESCRIPTION:
All employees at YKHC will be invited to complete an online survey that took approximately 10-15 minutes to complete. All employees will receive information via email, which includes an overview of the project, information regarding privacy and consent, and a link to the survey. Those who wish to do so were able to print a copy of the information for their reference. Employees who wish to participate did so by clicking on the survey link. Those who do not wish to participate could simply delete the email. Participants will be given two weeks to complete the online survey. Individuals who do not respond within the first week, will be sent an automated email reminder. All employees who participate will received a small incentive (approximately $10 in value).

ELIGIBILITY:
Inclusion Criteria:

* YKHC employee
* aged 18 years or older
* provides consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees at a health corporation in Western Alaska
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
current tobacco use | 7 days

IPD SHARING:
Plan to Share IPD: Yes